CLINICAL TRIAL: NCT04108390
Title: Effectiveness of Gluteus Medius Dry Needling in Patients With Chronic Ankle Instability
Brief Title: Gluteus Medius Dry Needling and Ankle Instability
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, Carlos Romero Morales, Principal Investigator, Universidad Europea de Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CIPI/19/012
Record Dates: First submitted 2019-09-26; First posted 2019-09-30 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Chronic Instability of Joint; Trigger Point Pain, Myofascial
Keywords: ankle; dry needling; trigger point
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Dry Needling; Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Individuals for this group will be treat with a dry needling intervention at the gluteus medius trigger point.
  Interventions: Other: Dry needling
- Control group (Active Comparator): Individuals for this group will be treat with a dry needling technique at 1,5 cm from the trigger point (not in the trigger point).
  Interventions: Other: Dry needling

INTERVENTIONS:
Other: Dry needling — For this intervention, the physiotherapist will be placed a needle in the gluteus medius trigger point from 8 to 15 times.
  Other Names: Manual Therapy

SUMMARY:
Randomized clinical trial in individuals with chronic ankle instability. Main outcomes were as follows: pain intensity, pressure pain threshold, lower limb balance and range of motion. The sample will be divided in two groups: 1) dry needling at the gluteus medius trigger point (intervention). 2) dry needling 1,5 cm from the gluteus medius trigger point (control).

DETAILED DESCRIPTION:
Inclusion criteria will be: individuals with chronic ankle instability, 20 to 50 years old. Exclusion criteria: any lower limb disease, fractures, infections, pregnancy, received any treatment in the previous 3 months.

Initially, the base measurements were as follows: paint intensity, pressure pain threshold at the gluteus medius trigger point, ankle range of motion and balance of the lower limb.

Once baseline measurements will be taken, the same evaluations will be performed at 4 weeks from the start.

ELIGIBILITY:
Inclusion Criteria:

* individuals with chronic ankle instability, 20 to 50 years old.

Exclusion Criteria:

* any lower limb disease, fractures, infections, pregnancy, received any treatment in the previous 3 months.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-03-25 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 1 day
  Individuals reported the pain intensity with the Visual Analogue Scale (VAS scale). The minimum and maximum scores were 0 (no pain) 100 (the worst pain). There was no sub-scales.
Pain pressure threshold | 1 day
  Pain pressure threshold were recorded with a pressure algometer. Evaluator press the trigger point with the algometer until the patient feel pain. The outcome will be recorder and expressed in kg/cm2

SECONDARY OUTCOMES:
Range of motion | 1 day
  Assess the ankle range of motion with a goniometer.
Balance | 1 day
  Assess the lower limb balance with the star excursion balance test

CONTACTS AND LOCATIONS:
Locations (1):
- Fiom clinic, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes